CLINICAL TRIAL: NCT00001002
Title: Intermittent Foscarnet Therapy for Human Immunodeficiency Virus Infection in Patients Receiving Long-Term Zidovudine Therapy
Brief Title: A Study of Foscarnet in the Treatment of HIV Infection in Patients Who Have Taken Zidovudine for a Long Time
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 053; 11027 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Foscarnet; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine; Foscarnet

INTERVENTIONS:
Drug: Zidovudine
Drug: Foscarnet sodium

SUMMARY:
To study the toxicity, pharmacokinetics, and antiretroviral effectiveness of combined oral zidovudine (AZT) and intermittent intravenous foscarnet therapy in stable AIDS or AIDS related complex (ARC) patients who have already received AZT for 8 - 52 weeks.

It is hypothesized that the maximum AZT antiretroviral effect, which occurs at 8 weeks of therapy, will be enhanced by 2 weeks of foscarnet treatment, given at the same time by intermittent intravenous infusion. In addition, the further lowering of serum p24 antigen concentration that should occur during combined therapy might continue when oral AZT therapy is continued without foscarnet.

DETAILED DESCRIPTION:
It is hypothesized that the maximum AZT antiretroviral effect, which occurs at 8 weeks of therapy, will be enhanced by 2 weeks of foscarnet treatment, given at the same time by intermittent intravenous infusion. In addition, the further lowering of serum p24 antigen concentration that should occur during combined therapy might continue when oral AZT therapy is continued without foscarnet.

There is a 4-week prestudy monitoring period during which AZT alone is administered on an outpatient basis, followed by a 2-week study period during which both intravenous foscarnet and oral AZT are administered in the hospital. During the subsequent 6-month follow-up period, oral AZT is administered and patients receive clinical evaluations. AZT is held for 48 hours on days before hospitalization and for 24 hours at the end of the hospitalization.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Medication necessary for the patient's welfare at the discretion of the investigator.

Patients must have the following:

* Received zidovudine (AZT) 200 mg every 4 hours (q4h) continuously for 8 - 16 weeks without Grade 3 or higher toxicity.
* Detectable p24 antigen in serum on at least 2 occasions during the prestudy period. All serum p24 antigen concentrations measured during the prestudy period must be at least twice the concentration cutoff value of the assay.
* Capability of giving informed consent.
* Per amendment of 890721, patients must enter the study period by September 30, 1989.

Exclusion Criteria

Co-existing Condition:

Patients with the following will be excluded:

* A history of hypersensitivity reaction to foscarnet or zidovudine (AZT).
* History of Grade 3 or 4 toxicity with AZT.
* Current Grade 2 or higher AZT toxicity.
* Osteomalacia, neoplasm metastatic to bone, or other known bone disease.
* Active opportunistic infection requiring myelosuppressive or nephrotoxic therapy.

Concurrent Medication:

Excluded:

* Antimetabolites.
* Immunomodulators.
* Nephrotoxins.
* Antiviral therapy.
* Myelosuppressive or nephrotoxic therapy.
* Acetaminophen.

Patients with the following will be excluded:

* A history of hypersensitivity reaction to foscarnet or zidovudine (AZT).
* History of Grade 3 or 4 toxicity with AZT.
* Current Grade 2 or higher AZT toxicity.
* Osteomalacia, neoplasm metastatic to bone, or other known bone disease.
* Active opportunistic infection requiring myelosuppressive or nephrotoxic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Study Completion 1991-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacobson MA, Study Chair
Locations (2):
- United States (2):
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - Unc Aids Crs, Chapel Hill, North Carolina

REFERENCES:
- [Background] Jacobsen MA, van der Horst C, Causey DM, Dehlinger M, Hafner R, Mills J. In vivo additive antiretroviral effect of combined zidovudine and foscarnet therapy for human immunodeficiency virus infection (ACTG Protocol 053). J Infect Dis. 1991 Jun;163(6):1219-22. doi: 10.1093/infdis/163.6.1219. PMID 1828075
- [Background] Aweeka FT, Gambertoglio JG, van der Horst C, Raasch R, Jacobson MA. Pharmacokinetics of concomitantly administered foscarnet and zidovudine for treatment of human immunodeficiency virus infection (AIDS Clinical Trials Group protocol 053). Antimicrob Agents Chemother. 1992 Aug;36(8):1773-8. doi: 10.1128/AAC.36.8.1773. PMID 1416864